CLINICAL TRIAL: NCT02864212
Title: Development of a Methodology to Design a High Order Sliding Mode Controller for Drug Dosage
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Other Study IDs: R-2014-785-063
Record Dates: First submitted 2016-07-29; First posted 2016-08-11 (Estimated); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Diabetes; Hypertension; Anesthesia
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Glucose monitoring: Glucose will be monitor in patients using fast-acting insulin.
- Depth of anesthesia monitoring: Depth of anesthesia will be monitor in patients undergoing cardiac surgery.
- Blood pressure monitoring: Invasive blood pressure will be monitor in patients undergoing cardiac surgery.

SUMMARY:
The aim of this observational study is to create a data base to extract feature of fast-acting drugs that can be monitor in real time to design control strategies based on high order sliding mode controller to create a robust drug infusion system.

DETAILED DESCRIPTION:
The aim of this observational study is to create a database to extract feature of fast-acting drugs that can be monitor in real time to design control strategies based on high order sliding mode controller to create a robust drug infusion system.

The observed drugs in this study are fast acting insulin, propofol and sodium nitroprusside.

The effect of insulin will be measured by a continuous glucose monitor, the effect of propofol by a bispectral index monitor and the the effect of sodium nitroprusside by a invasive blood pressure monitor.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I, II, II

Exclusion Criteria:

* Impossibility to measure depth of anesthesia or invasive blood pressure. Impossibility of using glucose monitor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients scheduled for surgery in the Cardiology Hospital CMNSXXI or treated with fast-acting insulin in the Cardiology Hospital CMNSXXI
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Glucose | Every 5 minutes during 3 days.
  The glucose will be measured by a continuous glucose monitor. For the group of patients for diabetes.
  Note: This protocol has three primary outputs because its objective is to create a database of each output to analyze the response to the associated drug (insulin, propofol and sodium nitroprusside.
Bispectral Index | Every second during surgery
  Depth of anesthesia will be measured by a Bispectral Index monitor.
Invasive blood pressure | Every 5 minutes during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ana Gallardo, Dr, Principal Investigator — Investigator
Locations (1):
- Unidad de Investigación Médica en Enfermedades Metabólicas IMSS, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided